CLINICAL TRIAL: NCT05090592
Title: Influence of Corneal Biomechanical Properties on Myopia Reduction and Axial Elongation in Children Using Orthokeratology and 0.01% Atropine
Brief Title: Influence of Corneal Biomechanical Properties on Myopia Control
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Buddhist TCGH
Record Dates: First submitted 2021-09-07; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- myopic children: Myopic children use overnight orthokeratology or 0.01% atropine eye drop per night for myopia control
  Interventions: Device: orthokeratology; Drug: 0.01 atropine

INTERVENTIONS:
Device: orthokeratology — orthokeratology wearing for myopia control
Drug: 0.01 atropine — 0.01% atropine eye drop prevent myopic progression

SUMMARY:
to analyze the changes in corneal biomechanics of myopic children with different treatment (low concentration atropine eye drops and orthokeratology) and explore the possible mechanism of myopia control

DETAILED DESCRIPTION:
High myopia is accompanied by excessive growth of eyeball, which leads to many complications. Myopia control is a great concern of the government and ophthalmologists worldwide.

Atropine eye drops is used clinically to control the progression of myopia. In recent years, low dose Atropine eye drops (0.01%, 0.05% and 0.1%) have been proven to be effective in slowing growth of eyeball. With less negative effects, these eye drops have been widely used for school children in Taiwan. Orthokeratology is another effective tool to control myopia, and long-term wearing of Ortho-k lens can inhibit the speed of eyeball growth, it is the most useful optical treatment for myopia control.

The Corvis® ST is a combination of an air pulse tonometer with an ultra-high-speed Scheimpflug camera. The movement of the cornea is mainly influenced by three factors which can be measured by the instrument:

Intraocular pressure (IOP)，biomechanical properties of the cornea and corneal thickness. The relationship between adult corneal biomechanics and refractive error has been noted in recent years. Previous studies pointed out that corneal biomechanics analyzer (Corvis ST) can measure the deformation process of the cornea and the biomechanics parameters. These literature found that the corneas of myopic patients， esp. high myopic, have larger corneal deformation in biomechanics analysis and revealed that the corneal stiffness of myopia patients was lower. There are still few discussions about the effect of orthokeratology on corneal biomechanics and there is no research focused on the change of corneal biomechanics of low-concentration atropine user which is worthy of our further exploration.

In this study, the investigators hope to analyze the changes in corneal biomechanics of myopic children with different treatment (low concentration atropine eye drops and orthokeratology) and explore the possible mechanism of myopia control.

ELIGIBILITY:
Inclusion Criteria:

* myopia (<-1D)
* received Orthokeratology or 0.01% atropine for myopia control
* regular follow-up

Exclusion Criteria:

* ocular surface disease( dry eye, keratoconus..)
* allergy to orthokeratology or atropine
* received eye surgery

  * strabismus
  * premature birth

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We enroll the clinical patient who recieved orthokeratology or 0.01% atropine for myopia control. Age limits was 8 to 20 year-old. The purpose and process were carefully addressed to the subjects and their guardians who signed an informed consent form before commencing this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of the intraocular pressure in myopic children with different treatment | from the date of starting treatment, the IOP was measured 1 week, 1month and every 3 months up to 24 months.
  the investigators measure the intraocular pressure(IOP, mmHg) of myopic children with different treatment (low concentration atropine eye drops and orthokeratology)
changes of the visual acuity in myopic children with different treatment | from the date of starting treatment, the visual acuity was measured 1 week, 1month and every 3 months up to 24 months.
  the investigators measure the visual acuity of myopic children with different treatment (low concentration atropine eye drops and orthokeratology).
changes of the central corneal thickness in myopic children with different treatment | from the date of starting treatment, the central corneal thickness was measured 1 week, 1month and every 3 months up to 24 months.
  the the investigators measure the central corneal thickness(CCT, micrometer, ㎛) of myopic children with different treatment (low concentration atropine eye drops and orthokeratology) by Corvis ST machine
changes of the corneal biomechanics index in myopic children with different treatment | from the date of starting treatment, the corneal biomechanics index was measured 1 week, 1month and every 3 months up to 24 months.
  the the investigators measure the corneal biomechanics index (CBI) of myopic children with different treatment (low concentration atropine eye drops and orthokeratology) by Corvis ST machine
changes of the stress-strain index in myopic children with different treatment | from the date of starting treatment, the stress-strain index (SSI) was measured 1 week, 1month and every 3 months up to 24 months.
  the the investigators measure the stress-strain index (SSI) of myopic children with different treatment (low concentration atropine eye drops and orthokeratology) by Corvis ST machine

SECONDARY OUTCOMES:
changes of axial length in myopic children with different treatment | from the date of starting treatment, the axial length was measured, then repeat measure were performed every 6 months up to 24 months
  the investigators measure the axial length(mm) of eyeball of myopic children with different treatment (low concentration atropine eye drops and orthokeratology).

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Jen Chiu, Doctor, Study Director — Tzu Chi genral hospital
Locations (1):
- Yu-Teng Lai, Yilan, Ilan County, Taiwan